CLINICAL TRIAL: NCT07226232
Title: A Multi-site Randomized Controlled Trial of Psilocybin for Treatment-Resistant Depression (TRD) in Veterans
Brief Title: Psilocybin Intervention for Veterans Overcoming Treatment-Resistant Depression
Acronym: PIVOT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBC-002-25S
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Major Depression
Keywords: depression; psilocybin; veterans; post-traumatic stress disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Enrolled participants who meet eligibility criteria and attend 3 preparatory visits with a psychological support facilitator will be randomized to either the control group or the intervention group in parallel until the primary endpoint at week 4 post randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only pharmacist will know the treatment assignment. All others are masked to treatment assignment.
  For the 1st of 2 dosing sessions, Veterans are randomized to receive one of two doses of psilocybin. One month later, participants return for a 2nd psilocybin dosing session in which all participants get the same dose of psilocybin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Psilocybin comparator dose
  Interventions: Drug: Psilocybin
- Intervention (Experimental): Psilocybin intervention dose
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin comparator dose
  Other Names: COMP360
  Arms: Control
Drug: Psilocybin — Psilocybin Intervention Dose
  Other Names: COMP360
  Arms: Intervention

SUMMARY:
The purpose of this multi-site randomized controlled trial is to evaluate the efficacy and risks of psilocybin for the treatment of depression in U.S. military Veterans with and without (±) concurrent posttraumatic stress disorder.

DETAILED DESCRIPTION:
Treatment-resistant depression (TRD) is a serious mental health problem in Veterans, frequently comorbid with post-traumatic stress disorder (PTSD), and in need of novel and effective treatments. Clinical studies have revealed antidepressant effects of psilocybin for depression in civilians, but less is known about its efficacy and safety in Veterans. Very limited data is available on the effects of psilocybin in the treatment of PTSD. Thus, it is important to evaluate the safety and efficacy of psilocybin in the treatment of TRD with and without PTSD among Veterans.

The purpose of this multi-site, double-blind, randomized controlled trial is to evaluate the efficacy and risks of psilocybin for the treatment of TRD in U.S. military Veterans with and without (±) concurrent PTSD. Eligible and consenting Veterans will two psilocybin dosing sessions along with preparation, administration, and integration psychological support provided by a facilitator. For the 1st psilocybin administration, participants will be randomized to one of two doses under blinded conditions. One month later, all participants will receive a 25mg dose at their 2nd psilocybin visit. Outcomes will be measured by an independent evaluator masked from all treatments at 2 and 4 weeks after each dosing session. Longer-term follow-up will be conducted over 6 months. Both expected and unanticipated adverse events will be collected by type, severity and relatedness to the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of the U.S. military who is English-speaking
* Signed informed consent and HIPAA
* Adults </= 75 years of age
* Meets DSM-5 criteria for current major depressive episode (MDE)
* MADRS >/= 20 at baseline
* Failure to respond satisfactorily to >/= 2 antidepressant treatments for >/= 8 weeks, including >/= 2 weeks at an adequate dose (>/= 50% of the FDA-approved uppermost dose) for major depression. Augmentation with a medication for depression (e.g., neuroleptics, lithium, levothyroxine) is considered a separate course of treatment.
* If applicable, concurrent & permitted antidepressants must be at stable doses for >/= 4 weeks prior to baseline (see allowed & prohibited medication list)
* Participants of child-bearing potential must have negative pregnancy test & agree to adhere to a medically acceptable method of birth control during the study
* Has a responsible adult who will provide transportation to the participant's home or place of lodging on the days of psilocybin administration

Exclusion Criteria:

Exclusion Criteria:

* Lifetime bipolar, schizophrenia spectrum, or other psychotic disorders
* First-degree relative with history of bipolar I, schizophrenia spectrum or other psychotic disorder
* Presence of psychotic symptoms (e.g., MDE with psychotic symptoms)
* Sedative-hypnotic, stimulant, inhalant and/or opioid use disorder within past 6 months (lifetime substance use disorder is allowed at the discretion of the LSI)
* Severe alcohol and/or cannabis use disorder within the past 6 months (mild or moderate alcohol and/or cannabis use is allowed at the discretion of the LSI)
* Lifetime hallucinogen persisting perception or hallucinogen use disorders
* Use of psilocybin, ayahuasca, mescaline, lysergic acid diethylamide (LSD), dimethyltryptamine (DMT), 5-Methoxy-N,N-dimethyltryptamine (5-MeO-DMT), peyote, or 3,4-methylenedioxymethamphetamine (MDMA) within past 6 months
* Participant agrees to not use psychedelics (listed above) during the study, except as prescribed by the study protocol
* Taking prohibited medication within 2 weeks of baseline (see allowed and prohibited concomitant medication list)
* History of severe traumatic brain injury (TBI)
* Diagnosis of dementia or related progressive neurocognitive disorder
* Suicidal ideation/behavior Type 4 or Type 5 intensity on C-SSRS within past 6 months of baseline
* Psychiatric inpatient treatment within past 3 months of baseline
* Treatment with electroconvulsive therapy, deep brain stimulation, vagus nerve stimulation, or transcranial magnetic stimulation within 3 months of baseline
* Implanted central nervous system device
* Treatment with evidence-based psychotherapy (EBP) for MDD or PTSD within 2 weeks prior to baseline. If receiving EBP therapy, he/she must complete treatment at least 2 weeks prior to baseline. Other forms of non-EBP psychotherapy for MDD or PTSD are allowed to continue during the study period.
* Pregnancy or lactation, or anticipated pregnancy or breastfeeding during the active treatment phase
* History of myocardial infarction, congestive heart failure, diabetic ketoacidosis, brain cancer, stroke and/or severe cardiac disease
* Clinically significant cardiac, pulmonary, renal, liver and/or other medical disease that, in the opinion of the investigator, may contraindicate the use of psilocybin, interfere with the interpretation of study results and/or constitute a health risk for the participant if they take part in the study
* Seizure disorder, except for seizures due to fever or withdrawal from a substance
* Clinically significant hypertension (>160/95 mmHg), hypotension (<90/60 mmHg) tachycardia (>100 bpm at rest), QTc prolongation (>450 msec men; >470 msec women) or clinically significant arrhythmia on ECG
* Clinically significant abnormal laboratory results on chemistry panel, liver function tests, complete blood count, and/or thyroid stimulating hormone
* Positive urine drug screen for illicit drugs of abuse (except for THC) at screening or baseline
* Prior allergic, adverse reaction or adverse experience to a psilocybin formulation
* Litigating for disability income for a mental disorder outside the VA compensation and pension process

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-12-02 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Rating Scale (MADRS) | 2 weeks
  10-item clinician-administered rating scale for depression. Scored 0 to 60; higher score indicates more severe symptomatology.

SECONDARY OUTCOMES:
Swiss Psychedelic Side Effects Inventory Overall Score | one day
  A clinician guided self-report form that has a list of effects pertaining to psychedelics; has the option to add other side effects (or expected effects) as desired and includes an open text field to provide additional details that are not captured in the inventory list. In addition to rating severity of the side effects, the SPSI captures impact, causality, timing and duration, and has a global rating on tolerability. Scoring: Calculate total scores for the number of side effects, severity, and impact by adding the relevant columns. Calculate total scores for the number of side effects, severity, and impact by adding the relevant columns. The overall score is calculated by subtracting total severity from total impact. The overall score represents the burden of side effects for that person within the specified timeframe.

OTHER OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 - Revised | one month
  A 30-item interview used to rate the past-month PTSD severity in those participants diagnosed with PTSD by CAPS-5-R at baseline. Higher score (0 to 200) indicates higher PTSD severity.
Hamilton Depression Rating Scale | two weeks
  A validated rater-administered measure of depression severity. The 17-item version yields a score of 0 to 50; higher score indicates more severe depression.
Patient Health Questionnaire 9 | two weeks
  A 9-item self-report measure designed to characterize severity of depression; has excellent psychometrics, total score range 0 to 27, higher = more severe.
PTSD Checklist for DSM-5 | one month
  A 20-item self-report of PTSD symptoms; score 0-80; higher=more severe. Only collected in those with PTSD diagnosis at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Lynne Davis, MD AB, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (5):
- United States (5):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and a data dictionary will be shared pending required IRB approval, and if needed, a Data Use Agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the conclusion of the study after a data repository has been made operational.
Access Criteria: De-identified data of those participants who signed informed consent, to include baseline demographics and clinical characteristics, primary outcome measure over time, treatment assignment, secondary safety outcomes, and exploratory outcomes. Data will be available for 6 years after the closure of the main study.